CLINICAL TRIAL: NCT02196688
Title: A Randomized, Double-blind, Placebo-controlled, Multicenter Phase II Trial to Compare the Efficacy and Safety of Fruquintinib Plus Best Supportive Care (BSC) Versus Placebo Plus BSC in Patients With Colorectal Cancer as 3rd or Above Therapy
Brief Title: Study of Fruquintinib in Patients With Metastatic Colorectal Cancer
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Hutchison Medipharma Limited (Industry)
Collaborators: Fudan University (Other); Sun Yat-sen University (Other)
Responsible Party: Sponsor
Organization: Hutchmed (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2012-013-00CH1
Record Dates: First submitted 2014-07-14; First posted 2014-07-22 (Estimated); Results first posted 2019-08-13 (Actual); Last update posted 2020-06-16 (Actual); Status verified 2020-06

CONDITIONS: Colorectal Cancer
Keywords: Colorectal cancer; Fruquintinib; 013
MeSH Terms: conditions — Colorectal Neoplasms | interventions — HMPL-013

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- treatment arm (Active Comparator): treatment arm- subjects will receive Fruquintinib 5mg orally, once daily (QD), plus BSC for 3 wks on/ 1 wk off. Patients will receive a cycles of 4 weeks of study treatment (1 cycle of study treatment includes 3 weeks of treatment and 1 week of drug discontinuation) or until the occurrence of progressive disease (PD), death, unacceptable toxicity, withdrawal of consent or other conditions that meet the end of treatment criteria.
  Interventions: Drug: fruquintinib
- control arm (Placebo Comparator): control arm- subjects will receive Fruquintinib placebo 5mg orally, once daily (QD), plus BSC for 3 wks on/ 1 wk off. Patients will receive a cycles of 4 weeks of study treatment (1 cycle of study treatment includes 3 weeks of treatment and 1 week of drug discontinuation) or until the occurrence of progressive disease (PD), death, unacceptable toxicity, withdrawal of consent or other conditions that meet the end of treatment criteria.
  Interventions: Drug: placebo

INTERVENTIONS:
Drug: fruquintinib — fruquintinib is a capsule in the form of 1mg and 5mg, orally, once daily, 3 weeks on/ 1 week off
  Other Names: HMPL-013
  Arms: treatment arm
Drug: placebo — Placebo is a capsule in the form of 1mg and 5mg, orally, once daily, 3 weeks on/ 1 week off
  Other Names: HMPL-013 placebo
  Arms: control arm

SUMMARY:
Fruquintinib administered at 5mg once daily in 4 weeks treatment cycle (three weeks on and one week off) was well tolerated and demonstrated encouraging preliminary clinical antitumor activity in patients with advanced Colorectal Cancer (CRC) in Phase Ib study.

This study is aimed to evaluate the efficacy and safety of Fruquintinib in the treatment of patients with metastatic CRC who have progressed after metastatic CRC second line or above standard chemotherapy.

DETAILED DESCRIPTION:
This is a randomized, double-blind, placebo-controlled, multicenter Phase II clinical trial to compare the efficacy and safety of Fruquintinib plus Best Supportive Care (BSC) versus placebo plus BSC in patients with metastatic colorectal cancer who have progressed after second-line or above standard chemotherapy.

After checking eligibility criteria, subjects will be randomized into Fruquintinib plus BSC group (treatment group) or placebo plus BSC group (control group) in a ration of 2:1.

Primary Efficacy Endpoint:

Progression free survival (PFS) (According to RECIST Version 1.1).

Secondary Efficacy Endpoints:

Objective Response Rate (ORR), Disease Control Rate (DCR), Overall Survival (OS).

Safety and tolerance will be evaluated by incidence, severity and outcomes of adverse events (AEs) and categorized by severity in accordance with the NCI common terminology criteria for adverse events (CTC AE) Version 4.0.

ELIGIBILITY:
Inclusion Criteria:

* ≥ 18 and ≤ 75 years of age , with ≥ 40 Kg
* Histological or cytological confirmed metastatic colorectal cancer
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-1
* Failed 2 or more lines of chemotherapy
* Adequate hepatic, renal, heart, and hematologic functions
* At least one measurable lesion (larger than 10 mm in diameter by spiral CT scan)
* Signed and dated informed consent.
* Willingness and ability to comply with scheduled visits, treatment plans, laboratory tests, and other study procedure

Exclusion Criteria:

* Pregnant or lactating women
* Any factors that influence the usage of oral administration
* Central nervous system (CNS) metastasis
* One of the following conditions: non-controlled hypertension, coronary artery disease, arrhythmia and heart failure
* Abuse of alcohol or drugs
* Less than 4 weeks from the last clinical trial - Previous treatment with VEGFR inhibition
* Disability of serious uncontrolled intercurrence infection
* Proteinuria ≥ 2+ (1.0g/24hr)
* Evidence or a history of bleeding tendency within two months of the enrollment, regardless of seriousness
* History of artery/venous thromboembolic events in 12 months, such as cerebral vascular accident (including transient ischemic attack) etc.
* History of acute myocardial infarction, acute coronary syndrome or coronary artery bypass graft (CABG) in 6 months
* Bone fracture or wounds that was not cured for a long time
* Coagulation dysfunction, hemorrhagic tendency or receiving anticoagulant therapy

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2014-04; Primary Completion 2015-04 (Actual); Study Completion 2015-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jin Li, MD, Principal Investigator — Fudan University
Locations (5):
- China (5):
  - Hutchison Medi Pharma Investigational Site, Beijing, Beijing Municipality
  - Hutchison Medi Pharma Investigational Site, Guangzhou, Guangdong
  - Hutchison Medi Pharma, Harbin, Heilongjiang
  - Hutchison Medi Pharma Investigational Site, Hangzhou, Zhejiang
  - Hutchison Medi Pharma Investigational Site, Shanghai

REFERENCES:
- [Result] Xu RH, Li J, Bai Y, Xu J, Liu T, Shen L, Wang L, Pan H, Cao J, Zhang D, Fan S, Hua Y, Su W. Safety and efficacy of fruquintinib in patients with previously treated metastatic colorectal cancer: a phase Ib study and a randomized double-blind phase II study. J Hematol Oncol. 2017 Jan 19;10(1):22. doi: 10.1186/s13045-016-0384-9. PMID 28103904

RESULTS

PARTICIPANT FLOW:
Groups:
- Treatment Arm: treatment arm- subjects will receive Fruquintinib 5mg orally, Once Daily (QD), plus Best Supportive Care (BSC) for 3 wks on/ 1 wk off. Patients will receive a cycles of 4 weeks of study treatment (1 cycle of study treatment includes 3 weeks of treatment and 1 week of drug discontinuation) or until the occurrence of progressive disease (PD), death, unacceptable toxicity, withdrawal of consent or other conditions that meet the end of treatment criteria.
  fruquintinib: fruquintinib is a capsule in the form of 1mg and 5mg, orally, once daily, 3 weeks on/ 1 week off
- Control Arm: control arm- subjects will receive Fruquintinib placebo 5mg orally, Once Daily (QD), plus Best Supportive Care (BSC) for 3 wks on/ 1 wk off. Patients will receive a cycles of 4 weeks of study treatment (1 cycle of study treatment includes 3 weeks of treatment and 1 week of drug discontinuation) or until the occurrence of progressive disease (PD), death, unacceptable toxicity, withdrawal of consent or other conditions that meet the end of treatment criteria.
  placebo: Placebo is a capsule in the form of 1mg and 5mg, orally, once daily, 3 weeks on/ 1 week off
Period: Overall Study
Arm/Group | Treatment Arm | Control Arm
Started | 47 | 24
Completed | 40 | 23
Not Completed | 7 | 1

BASELINE CHARACTERISTICS:
Groups:
- Treatment Arm: treatment arm- subjects will receive Fruquintinib 5mg orally, QD, plus BSC for 3 wks on/ 1 wk off. Patients will receive a cycles of 4 weeks of study treatment (1 cycle of study treatment includes 3 weeks of treatment and 1 week of drug discontinuation) or until the occurrence of progressive disease (PD), death, unacceptable toxicity, withdrawal of consent or other conditions that meet the end of treatment criteria.
  fruquintinib: fruquintinib is a capsule in the form of 1mg and 5mg, orally, once daily, 3 weeks on/ 1 week off
- Control Arm: control arm- subjects will receive Fruquintinib placebo 5mg orally, QD, plus BSC for 3 wks on/ 1 wk off. Patients will receive a cycles of 4 weeks of study treatment (1 cycle of study treatment includes 3 weeks of treatment and 1 week of drug discontinuation) or until the occurrence of progressive disease (PD), death, unacceptable toxicity, withdrawal of consent or other conditions that meet the end of treatment criteria.
  placebo: Placebo is a capsule in the form of 1mg and 5mg, orally, once daily, 3 weeks on/ 1 week off
- Total: Total of all reporting groups
Arm/Group | Treatment Arm | Control Arm | Total
Number analyzed (Participants) | 47 | 24 | 71
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 41 | 20 | 61
  >=65 years | 6 | 4 | 10
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 7 | 19
  Male | 35 | 17 | 52
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 47 | 24 | 71
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 0 | 0 | 0
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  ETHNICITY: HAN | 47 | 24 | 71
  ETHNICITY: NOT HAN | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  China | 47 | 24 | 71

OUTCOME MEASURES:

1. Primary Outcome: Progression Free Survival (PFS)
Description: PFS refers to the time interval between the randomization date and the initial record of PD or date of death, whichever is earlier. The presence of PD shall be determined in accordance with the result of the evaluation performed by the investigator, using with RECIST v1.1 criteria. The date of final tumor evaluation will be used as the censoring date for subjects who have not presented with disease progression or death by that date. The date of randomization will be used as the censoring date for subjects which have no death and post-baseline tumor evaluation. If a subject has no post-baseline tumor evaluation but recorded as dead, death will be count as PFS event.
Time Frame: From randomization until the date of first documented progression or date of death from any cause, whichever came first.
Population: The intention-to-treat set will contain all subjects in the Randomized set (RND) set subjects will be classified according to randomized treatment. The intent-to-treat principle is preserved. The Intention to Treat (ITT) will be used for analyses of PFS, OS, ORR and DCR.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 47 | 24
months | 4.731 [2.858 to 5.585] | 0.986 [0.953 to 1.577]

2. Secondary Outcome: Objective Response Rate (ORR)
Description: The ORR is defined as the rate of complete response (CR) or partial response (PR) as the best overall response (BOR), based on evaluation of target lesions and non-target lesions with corroborant radiological method and determined by RECIST v1.1, for the ITT set of response evaluable subjects. Subjects who have no post-baseline tumor evaluation shall be regarded as subjects without ORR. Subjects who qualify for evaluation of CR or PR should have at least one available lesion for measurement with RECIST v1.1.
Time Frame: From randomization up to progressive disease or end of treatment (EOT) due to any cause.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 47 | 24
Participants | 1 | 0

3. Secondary Outcome: Disease Control Rate (DCR)
Description: The DCR is defined as the rate of corroborant CR, PR and stable disease (SD) as the BOR, based on evaluation of target lesions and non-target lesions with corroborant radiological method and determined according to RECIST v1.1, for the ITT set of response evaluable subjects.
Time Frame: From randomization up to progressive disease or EOT due to any cause.
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 47 | 24
Participants | 32 | 5

4. Secondary Outcome: Over Survival (OS)
Description: The OS refers to the time interval between the randomization date and the date of death (any cause). The final known date of survival will be used as the censoring date for subjects that have not been reported to have died by the time of analysis.
Time Frame: From randomization until death due to any cause.
Measure: Median (95% Confidence Interval); unit: months
Arm/Group | Treatment Arm | Control Arm
Number analyzed (Participants) | 47 | 24
months | 7.721 [6.899 to 10.283] | 5.520 [3.614 to 11.302]

ADVERSE EVENTS:
Time Frame: Adverse event (AE) should be collected from first dose to 30 days after EOT. AEs and laboratory abnormalities that could not be restored or unexplained needed to be collected till recovery or until they could be explained. Serious adverse event (SAE) was collected from informed consent. Only SAEs related to the study drugs should be collected until 30 days after the last dose.
Arm/Group | Treatment Arm | Control Arm
All-Cause Mortality (participants affected / at risk) | 38/47 | 19/24
Serious Adverse Events (participants affected / at risk) | 12/47 | 5/24
Other Adverse Events (participants affected / at risk) | 47/47 | 20/24
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=47) | Control Arm (N=24)
Hypertension (Vascular disorders) | 3 | 0
Embolism arterial (Vascular disorders) | 1 | 0
Superior vena cava syndrome (Vascular disorders) | 1 | 0
Obstruction intestinal (Gastrointestinal disorders) | 2 | 0
Pancreatitis acute (Gastrointestinal disorders) | 1 | 0
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0
Functional ileus (Gastrointestinal disorders) | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 1 | 0
Hepatic damage (Hepatobiliary disorders) | 1 | 0
Jaundice cholestatic (Hepatobiliary disorders) | 1 | 0
Pyrexia (General disorders) | 2 | 0
Sudden death (General disorders) | 0 | 1
Blood bilirubin increased (Investigations) | 2 | 0
Platelet count decreased (General disorders) | 0 | 1
Dyskinesia (Nervous system disorders) | 1 | 0
Hepatic coma (Nervous system disorders) | 0 | 1
Haemoptysis (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Muscle weakness (Musculoskeletal and connective tissue disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment Arm (N=47) | Control Arm (N=24)
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 15 | 3
BLOOD THYROID STIMULATING HORMONE INCREASED (Investigations) | 11 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 9 | 1
BLOOD BILIRUBIN INCREASED (Investigations) | 9 | 3
OCCULT BLOOD POSITIVE (Investigations) | 8 | 3
PLATELET COUNT DECREASED (Investigations) | 8 | 1
BLOOD ALKALINE PHOSPHATASE (Investigations) | 7 | 3
WHITE BLOOD CELL COUNT DECREASED (Investigations) | 6 | 0
ELECTROCARDIOGRAM T WAVE AMPLITUDE DECREASED (Investigations) | 5 | 0
NEUTROPHIL COUNT DECREASED (Investigations) | 5 | 0
WEIGHT DECREASED (Investigations) | 5 | 0
BLOOD PRESSURE INCREASED (Investigations) | 4 | 0
BLOOD URINE PRESENT (Investigations) | 3 | 1
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 0 | 2
BLOOD POTASSIUM DECREASED (Investigations) | 0 | 2
HAEMOGLOBIN DECREASED (Investigations) | 0 | 3
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 30 | 2
NAIL DISCOLOURATION (Skin and subcutaneous tissue disorders) | 9 | 0
RASH (Skin and subcutaneous tissue disorders) | 7 | 0
DERMATITIS ACNEIFORM (Skin and subcutaneous tissue disorders) | 5 | 2
RASH MACULO-PAPULAR (Skin and subcutaneous tissue disorders) | 3 | 0
FATIGUE (General disorders) | 15 | 2
MALAISE (General disorders) | 10 | 2
PYREXIA (General disorders) | 8 | 3
ASTHENIA (General disorders) | 5 | 2
INFLUENZA LIKE ILLNESS (General disorders) | 3 | 1
DIARRHOEA (Gastrointestinal disorders) | 15 | 3
STOMATITIS (Gastrointestinal disorders) | 12 | 1
CONSTIPATION (Gastrointestinal disorders) | 7 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 6 | 2
VOMITING (Gastrointestinal disorders) | 6 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 5 | 2
NAUSEA (Gastrointestinal disorders) | 5 | 2
ABDOMINAL DISTENSION (Gastrointestinal disorders) | 3 | 2
APHTHOUS STOMATITIS (Gastrointestinal disorders) | 3 | 0
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 25 | 2
COUGH (Respiratory, thoracic and mediastinal disorders) | 9 | 0
PROTEINURIA (Renal and urinary disorders) | 22 | 5
HAEMATURIA (Renal and urinary disorders) | 6 | 1
DECREASED APPETITE (Metabolism and nutrition disorders) | 14 | 4
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 8 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 4 | 0
HYPOKALAEMIA (Metabolism and nutrition disorders) | 4 | 0
HYPONATRAEMIA (Metabolism and nutrition disorders) | 2 | 2
HYPERTENSION (Vascular disorders) | 21 | 3
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 | 0
BACK PAIN (Musculoskeletal and connective tissue disorders) | 8 | 2
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 2
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 2 | 2
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 7 | 1
URINARY TRACT INFECTION (Infections and infestations) | 4 | 0
ANAEMIA (Blood and lymphatic system disorders) | 7 | 1
DIZZINESS (Nervous system disorders) | 3 | 0
TINNITUS (Ear and labyrinth disorders) | 5 | 0
HEPATIC PAIN (Hepatobiliary disorders) | 2 | 2
SINUS TACHYCARDIA (Cardiac disorders) | 3 | 1
HYPOTHYROIDISM (Endocrine disorders) | 3 | 0
INSOMNIA (Psychiatric disorders) | 3 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No